CLINICAL TRIAL: NCT06770309
Title: A Prospective, Double-blind, Randomized Controlled Clinical Study of Silkworm Pupa Powder Intervention in the Nutritional Status of Patients with Alzheimer's Disease
Brief Title: A Study of Silkworm Pupa Powder Intervention in the Nutritional Status of Patients with Alzheimer's Disease.
Acronym: AD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yanbu Ke (Other)
Responsible Party: Sponsor-Investigator, Yanbu Ke, The director of Hangzhou First People's Hospital(Hangzhou Geriatric Hospital), First People's Hospital of Hangzhou
Organization: First People's Hospital of Hangzhou (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: syyycanyongfen
Record Dates: First submitted 2024-12-29; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease (AD); Sarcopenia; Asthenia
Keywords: Alzheimer Disease; Sarcopenia; asthenia; nutritional status
MeSH Terms: conditions — Alzheimer Disease; Sarcopenia; Asthenia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Silkworm pupa powder, 2 times a day, two packets (12*2 g) each time, take with warm water, before meals, for three months
  Interventions: Dietary Supplement: Silkworm pupa powder
- Control group (Placebo Comparator): Placebo, 2 sachets (12*2 g) twice a day, with warm water, before meals, for three months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Silkworm pupa powder — Silkworm pupa powder, 2 times a day, two packets (12*2 g) each time, take with warm water, before meals, for three months
  Arms: Experimental group
Dietary Supplement: Placebo — Placebo, 2 sachets (12*2 g) twice a day, with warm water, before meals, for three months
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if silkworm pupa powder works to improve the nutritional status of Alzheimer's disease patients. The main questions it aims to answer are:

* Does silkworm pupa powder evaluate the effectiveness of silkworm pupae in improving sarcopenia, frailty and quality of life in AD patients?
* Does silkworm pupa powder improve cognitive function in AD patients?

Researchers will compare silkworm pupa powder to a placebo (a look-alike substance that contains no drug) to see if silkworm pupa powder works to improve the nutritional status of Alzheimer's disease patients.

Participants will:

* Take drug silkworm pupa powder or a placebo every day for 3 months.
* Visit the clinic once every 4 weeks for checkups and tests.
* Keep a diary of their daily consumption.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for dementia caused by AD as determined by the National Institute on Aging and the Alzheimer's Disease Association (NIA-AA) (2024);
2. Male or menopausal female (no fertility requirement), participants are 50-90 years old (inclusive) with primary school education or above;
3. The Mini Mental State Examination (MMSE) score for illiteracy is ≤ 17 points, primary school education is ≤ 20 points, secondary school education is ≤ 22 points, and university education is ≤ 23 points; CDR>2.0 points;;
4. 0 points< 40 points ≤ the ADL Rating Scale;
5. At the time of screening and enrollment, there was a nutritional risk score of ≥3 points (according to the NRS2002 Nutritional Risk Screening Form);
6. In good general condition, ECOG score ≤ 3 points;
7. If you are receiving approved Alzheimer's disease treatment, such as acetylcholinesterase inhibitors, GV-971, NMDA receptor antagonists, you must maintain a stable dose for at least 12 weeks before baseline, and the cognitive evaluation scale is stable. Participants who have not been treated for Alzheimer's disease may be enrolled. Unless otherwise noted, participants must maintain a stable dose of all other (i.e., non-Alzheimer's disease-related) permitted concomitant medications for at least 4 weeks prior to baseline;
8. The investigator confirms that the subject has a stable and reliable caregiver;
9. You voluntarily participate in this clinical research, fully understand and be informed about the study, and sign the informed consent form (ICF).； Willing to follow and able to complete all trial procedures. If the participant lacks the capacity to consent in the opinion of the investigator, the participant's consent shall be obtained as required by local laws, regulations, and customs. (or signed by the patient's caregiver with the authorization of the patient's guardian) during the study to agree to provide peripheral blood, feces, urine, samples for biomarker analysis.

Exclusion Criteria:

1. Dementia caused by the following reasons: vascular dementia, central nervous system infection (such as AIDS, syphilis, etc.), Huntington's disease and Parkinson's disease, dementia with Lewy bodies, traumatic brain dementia, other physical and chemical factors (such as drug poisoning, alcohol poisoning, carbon monoxide poisoning, etc.), important physical diseases ( Such as hepatic encephalopathy, pulmonary encephalopathy, hypoxic encephalopathy, etc.), intracranial mass lesions (such as subdural hematoma, brain tumors), endocrine system lesions (such as thyroid disease, adrenal gland disease) as well as dementia caused by vitamins or any other cause;
2. Patients with other autoimmune diseases, such as multiple sclerosis, polymyositis, myasthenia gravis, Guillain-Barré syndrome, ankylosing spondylitis, rheumatoid arthritis, systemic lupus erythematosus, vitiligo, etc.;
3. Severe renal insufficiency: creatinine clearance rate < 30mL/min (Cockcroft-Gault formula).or other known severe renal insufficiency disease; Severe hepatic impairment: ALT or AST > 10 times the upper limit of normal, or other known liver diseases such as acute and chronic active hepatitis, liver cirrhosis, etc.; During the screening period, patients with acute myocardial infarction or interventional therapy in the past 6 months, and heart failure (patients classified as grade III-IV according to NYHA); Patients with other serious primary diseases of the nervous system, heart, pulmonary, hematopoietic system or endocrine system and psychiatric disorders;
4. Those who suspect or have a history of alcohol or drug abuse;
5. Estimated survival ≤ 3 months;
6. Pregnant women or lactating women, subjects of childbearing age (including male subjects with heterosexual intercourse and their female partners of childbearing potential) who have pregnancy plans or are unwilling to take effective contraceptive measures from the beginning of screening to 3 months after discontinuation;
7. Those who are allergic to the ingredients of known test supplies
8. Participated in other drug clinical trials within 30 days before screening, or are participating in other clinical trials;
9. Patients with other serious physical or psychiatric diseases or laboratory abnormalities that may increase the risk of participating in the study and who are considered by the investigator to be unsuitable for participating in this study
10. Clinically severe mental disorder or psychiatric symptoms;
11. Mini-Mental State Assessment Scale (MMSE) score > 26 points;
12. Activity of daily living ability (ADL) rating scale > 40 points
13. Patients with abnormally elevated tumor markers or a history of tumor or no clear tumor;
14. Those who are at serious risk of suicide;
15. Patients who are intolerant or allergic to the drugs used in this study;
16. Clinically significant cardiovascular or cerebrovascular disease requiring treatment within 1 6 months or current diagnosis within 2 months;
17. Use of antibiotics: a. Use of antibiotics for more than 10 consecutive days in the 12 weeks prior to baseline; b. Subjects are expected to be treated with antibiotics for more than 10 days; Any other medical condition (e.g., cardiac, respiratory, renal disease, gastrointestinal disease that may affect absorption, such as gastric cancer, gastric bypass, or recurrent diarrhea) that is not stable and adequately controlled, or that, in the opinion of the investigator, may affect the safety of the participant or interfere with study assessments;
18. Any other clinically significant abnormality in physical examination, vital signs, laboratory tests, or ECG that, in the opinion of the investigator, requires further investigation or treatment, or may interfere with study procedures or safety;
19. Participants with bleeding disorders that are not adequately controlled (including platelet count< 50*10^9/L or international normalized ratio [INR]>1.5 for participants who did not receive anticoagulation therapy, e.g., warfarin);
20. Other circumstances that the researcher deems inappropriate to participate in this study.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | The 4th 、8th and 12th week after taking Silkworm
  Take blood testing and detect hemoglobin levels
Albumin | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Detect blood albumin levels
Serum prealbumin | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Detect serum prealbumin levels
25-hydroxyvitamin D | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Detect blood 25-hydroxyvitamin D levels
Alkaline phosphatase | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Detect blood alkaline phosphatase levels
Parathyroid hormone | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Detect parathyroid hormone levels
Calcitonin | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Detect calcitonin levels
Whole abdominal Computerized tomography (CT) scan | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Take the whole abdominal CT scan
Diagnostic criteria of the 2019 Asian Sarcopenia Working Group | The 4th 、8th and 12th week after taking Silkworm pupa powder.
  Evaluate sarcopenia again

SECONDARY OUTCOMES:
Mini-mental State Examination（MMSE） Scale | The 4th、8th and 12th week after taking placebo.
  Take the MMSE Scale again
Clinical Dementia Rating（CDR） Scale | The 4th 、8th and 12th week after taking placebo.
  Take the CDR Scale again
Eastern Cooperative Oncology Group Score | The 4th 、8th and 12th week after taking placebo.
  Take the ECOG Score again
Head Magnetic Resonance Scan | The 4th 、8th and 12th week after taking placebo.
  Take Head MR again
Amyloid β-protein（Aβ） | The 4th 、8th and 12th week after taking placebo.
  Detect the blood Amyloid β-protein levels, include Aβ42、Aβ40、Aβ40/42
Phosphorylated microtubule-associated protein Tau（P-Tau） | The 4th 、8th and 12th week after taking placebo.
  Detect the Phosphorylated microtubule-associated protein Tau levels, include P-tau181、P-tau 217

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Our research is in the exploratory stage and it is not yet clear what results will be obtained.